CLINICAL TRIAL: NCT04541901
Title: Effects of Post Exercise Massage and Cold-water Immersion on Movement Variability After Fatigue in Swimmers: a Randomized Controlled Clinical Trial
Brief Title: Massage and Cold Water Immersion on Movement Variability After Fatigue in Swimmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Flávia Carvalho (Other)
Collaborators: Universidade Estadual Paulista JÃºlio de Mesquita Filho (Unknown); São Paulo State University (Other)
Responsible Party: Sponsor-Investigator, Flávia Carvalho, MSc, São Paulo State University
Organization: São Paulo State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ECD001; 2020/11146-0 (Other Grant/Funding Number: São Paulo Research Foundation); 001 (Other Grant/Funding Number: Coordination of Superior Level Staff Improvement)
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Movement Disorders; Muscle Tone; Perceived Exertion
Keywords: Swimming; Massage; Cryotherapy; movement variability
MeSH Terms: conditions — Movement Disorders | interventions — Massage

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Massage (Experimental): 12 minutes of effleurage and petrissage on the upper limbs administered after fatiguing exercise in the swimming pool
  Interventions: Other: Massage
- Cold-water immersion (Experimental): 12 minutes of cold-water immersion at the shoulder level with water temperature between 11 to 15°C
  Interventions: Other: Cold water immersion
- Control (No Intervention): 12 minutes of rest. The athletes are free to sit or walk around the place but are advised to refrain from exercise in and out of the pool.

INTERVENTIONS:
Other: Massage — 12 minutes of effleurage and petrissage on the upper limbs
  Arms: Massage
Other: Cold water immersion — 12 minutes of cold water immersion at the shoulder level with water temperature between 11 to 15°C
  Arms: Cold-water immersion

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of post-exercise massage and cold-water immersion compared to control in young elite swimmers. The main questions it aims to answer are:

* Is post-exercise techniques effective for recovery of the movement variability, , myotonometric, ergometric and perceptive parameters after fatigue?
* Can neuromuscular fatigue protocols impair movement variability, myotonometric, ergometric and perceptive parameters?
* What tests are reliable to assess different aspects of swimmers' recovery?

Researchers will compare massage and cold-water immersion to control and to each other to see if recovery is antecipated. They will also compare an in-water and an out-of-water fatigue protocol to see if they are effective and can be used in different settings.

Participants will:

* Perform test and retest sessions to assess movement variability, myotonometric, ergometric and perceptive parameters.
* Perform an in-water fatigue protocol consisting of 8x100m front-crawl sprints
* Receive three recovery strategies in a randomized order (massage, cold-water immersion and control (i.e. rest)
* Answer a questionnaire regarding ther beliefs and preferences for recovery.

ELIGIBILITY:
Inclusion Criteria:

* male and female athletes
* between 15 and 30 years old
* no injury over the last month (any complaint that prevented the athlete from training or compete at least once)

Exclusion Criteria:

* use of pain killers at least 24h before study participation

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Movement variability | From enrollment to the end of crossover treatments at 6 weeks
  Obtained from time series of biomechanical data expressed as degrees of shoulder and elbow flexion, and ergometric variables (i.e. pace, stroke frequency and average power) executed during a simulated out of water swim ergometric test to understand the impacts of fatigue on movement and explore changes during recovery. Measured at baseline, post-fatigue and post-interventions.
  Joint angles time series of shoulder and elbow flexion and ergometric variables were aggregated using mean, standard deviation and variation coefficients for data analyses.

SECONDARY OUTCOMES:
Swim-related perceptions | From enrollment to the end of crossover treatments at 6 weeks
  Self-reported ratings regarding physical and mental readiness for exercise, fatigue, vigor, somnolence, pain, and perception of effort and recovery, measured by a numerical rating scale ranging from 0 (nothing) to 10 (extreme). Measured at baseline, post-fatigue and post-interventions
Myotonometry | From enrollment to the end of crossover treatments at 6 weeks
  Muscle tone, stiffness and elasticity were assessed by the MyotonPRO. The equipment probe will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at 1: Deltoid; 2: Pectoralis Major; 3: Biceps brachii; 4: Upper Trapezius; 5: Latissimus dorsi; 7: Triceps. Values were deemed acceptable if there were less than 3% of variation between the impulses. Measured at baseline, post-fatigue and post-interventions.
Skin temperature | From week 4 to 6
  The temperature will be measured using an infrared thermographic camera, at the same points of myotonometry. Measured before and after the interventions.
Beliefs in the recovery techniques | Week 6
  Participants will be asked if they believe that massage, cold-water immersion and resting contribute to their recovery before and after the study
Preference | Week 6
  After the study the participants will be asked which of the interventions they preferred to received to recover from the fatiguing exercise
Sense of position | From enrollment to the end of crossover treatments at 6 weeks
  Participants will be asked to position their dominant upper limb at 90° which will be indicated by a target fixed on the wall 1 meter ahead of them. They will have 3 chances to point at the target and memorize the position. Afterwards, participants will have 3 chances to point at the target without vision (by blindfold). Measured at baseline, post-fatigue and post-interventions

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Pastre, Doctor, Study Director — University of São Paulo State, UNESP
Locations (1):
- Faculty of Science and Technology (UNESP), Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared because they belong to a competitive team and most of the participants have less than 18 years old